CLINICAL TRIAL: NCT01433211
Title: Relation Between Nutrition and Frailty in Community-dwelling Older Persons
Brief Title: Nutrition and Frailty in Older Persons
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Dorothee Volkert, Professor Dr., University of Erlangen-Nürnberg Medical School
Other Study IDs: IBA-2011(1)
Record Dates: First submitted 2011-09-07; First posted 2011-09-13 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Frailty
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No treatment

SUMMARY:
The purpose of this study is to investigate the association between nutrition and frailty in older community-living persons.

DETAILED DESCRIPTION:
Nutrition is regarded as an important etiologic factor in the development of frailty in older adults. To date the relation between nutrition and frailty is only poorly described.

Thus, it is the purpose of this study to investigate the association between different nutrition characteristics and frailty in older community-living persons.

206 volunteers aged 75 years or older were included in this cross-sectional study. Nutritional assessment included the Mini-Nutritional Assessment (MNA), a food-frequency questionnaire and a standardised three-day dietary record. Intake of energy and nutrients was calculated using the German nutrient database BLS II.2. Dietary patterns were described by different dietary scores. Frailty was defined according to Fried et al. based on the following criteria: weight loss, exhaustion, grip strength, walking speed and physical activity. In addition several standardised tests were performed to characterise physical performance (Timed Up & Go, repeated chair stands, balance tests).

The association between nutritional aspects and physical performance is evaluated in an explorative manner.

ELIGIBILITY:
Inclusion Criteria:

* age of 75 years and older
* living independently at home

Exclusion Criteria:

* acute illness
* cognitive impairment (Mini Mental State Examination ≥ 24 out of 30 points)

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Community-living persons aged 75 years or older
Sampling Method: Probability Sample
Enrollment: 206 (Actual)
Dates: Start 2009-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Frailty (according to Fried et al.) | 1 day
  Frailty is defined as the presence of at least 3 of the following criteria:
  * self-reported weight loss of more than 4.5 kg in the last year
  * exhaustion (self-reported feeling that everything was an effort or one could not get "going" > 2 times a week)
  * low grip strength (men ≤ 29-32 kg, women ≤ 17-21 kg depending on BMI),
  * low walking speed (> 6-7 sec/ 4.57 m, depending on gender and height)
  * low physical activity (men < 383 kcal/ week, women < 270 kcal/ week)

SECONDARY OUTCOMES:
Impaired physical performance (according to Guralnik et al.) | 1 day
  Impaired physical performance is definded as less than 9 points in the Short Physical Performance Battery (SPPB).
  Three physical performance tests (balance, walking speed and chair-rise) are performed in a standardised manner and rated with 0-4 points each. SPPB is the sum score of these three test resuslts with a maximum of 12 points indicating the best physical performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Biomedicine of Aging, University of Erlangen-Nürnberg, Nuremberg, Germany

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356